CLINICAL TRIAL: NCT06812182
Title: Effectiveness a Nurse Guided Enhanced Recovery Pathway on Postoperative Respiratory Tract Infection in Hepatico-Pancreatic -Biliary Surgery
Brief Title: Effect of Nurse Guided Enhanced Recovery Clinical Pathway on Respiratory Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Abd El-Khalek Mohammed Glala, lecturer, Assiut University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Screening
Other Study IDs: Enhanced recovery clinical
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Nurse's Role

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): All the patients admitted to surgical department during the period from early Augusts 2023until the end November 2023 matching the inclusion criteria for this study were included in the control group. The control group contained 30 patients with the same designed criteria. The control group received routine daily care of the hospital. For the control group, the two designed study tools used to assess the patients daily and detect the clinical outcomes of the patients [tool I and tool III] only.
- study group (Experimental): educational training sessions were provided to care providers including the purpose and the process of implementing the pathway for one week. Following the training thee researchers started to make recruitment and screen for the study group, the researchers received consent from administration to start the data for the study group. The oral and written consent from the patient was also done, to allow the researchers to observe, make daily assessment and manage the patients according to the designed clinical pathway.
  After completion of the recruitment and screening, all patients admitted to the surgical unit during the five months period from first December 2023 until the end of April 2024 were assessed and managed as study group. The study group also estimated 30 patients that met the inclusion criteria. For the study group, the three designed study tools used to assess the patients daily and detect the clinical outcomes of the patients [tool I, tool II and tool III]
  Interventions: Behavioral: nurse guided clinical pathway

INTERVENTIONS:
Behavioral: nurse guided clinical pathway — Educational training sessions were provided to care providers for one week. Pre-operative; counseling and education of patient for chest physiotherapy, using spirometry, bowel preparation, early mobilization and how to predict common complications with learning to cooperate with nurses. Emphasis on patients to co-operate postoperatively was strongly stressed in spite of the pain and weakness.
  Intra-operative: Optimal fluid management, short acting anesthetics, regional analgesia, opioids-sparing anesthesia, small incisions, avoiding drains, maintaining normothermia, venous thrombo-embolism [VTE] prophylaxis and antibiotic prophylaxis were routinely done.
  Post-operative: Early oral nutrition, optimal fluid management, multimodal non-opioid analgesia, postoperative nausea and vomiting PONV prophylaxis, stimulation of gut motility, early removal of catheters and drains, early mobilization, chest physiotherapy and using spirometry effectively.
  Arms: study group

SUMMARY:
Objectives: Evaluate the effect of a nurse guided enhanced recovery pathway on postoperative respiratory tract infection in Hepatico-Pancreatic -Biliary surgery [ pre-operative patient counselling for postoperative respiratory physiotherapy techniques and emphasis on perfect training]. Design: Quasi-experimental study. Setting: The study was conducted in surgical department, operation unit and intensive care unit at AlRajhy liver hospital. Subjects: Sixty patient undergoing hepatobiliary pancreatic surgeries. The sample was divided into two groups; control and study group (30patient each). The control started the first then the study group. Tools: Three tools were used. Tool I: Patient assessment sheet. Tool II: Clinical pathway protocol. Tool III: Clinical outcome evaluation. The control group received tools I and III only while study group received the three tools including clinical pathway protocol [tool II].

DETAILED DESCRIPTION:
: Sixty patient undergoing hepatobiliary pancreatic surgeries. The sample was divided into two groups; control and study group [30patient each]. The control started the first then the study group.

The sample size was calculated according to Epi Info 2000. A sample size was selected using a special formula based on prevalence of disease at a confidence interval of 95% and precision of (2%). The sample was increased by 10% to overcome problems related to non-responses and missing data. The power of study was 80%. Considering the following matching criteria age group, sex, diagnosis, comorbidity diseases.

The patients' inclusion criteria: Age 18-65 years old, able to communicate and Patients without vital failure [renal, hepatic, cardiac].

The patients' exclusion criteria: Past history of other organ cancer and patient refusal.

Tools:

Tool one; Patient assessment sheet:

This tool was developed by researchers based on related literature to assess the surgical patient[11]. It consisted of three parts Part1: it included socio-demographic data about the patients such as: age, gender, level of education, material status and clinical data such as patient diagnosis, past medical history, past surgical history, surgical procedure and type of anesthesia.

Part 2: Intra¬¬-operative data which included estimated blood loss, urine output, fluid and blood replacement, final balance, intraoperative complications, duration of anesthesia, duration of surgical procedure and duration of recovery.

Part 3: Post-operative assessment that included:

Physical assessment included anthropometric measurement [weight, height and body mass index] body mass index measured through dividing weight by kg on the square of height by m2, vital sign [temperature, pulse, respiration, blood pressure] Monitoring Signs of respiratory infection [cough, dyspnea, hypoxemia, tachypnea] and the need to oxygen therapy were also recorded besides monitoring arterial blood gases.

Tool two [the main research investigation] = named as clinical pathway protocol:

Clinical pathway for hepatobiliary pancreatic surgeries, this tool was developed by researchers after extensive review of related literatures and enhanced recovery after surgery pathway. The researchers used enhanced recovery after surgery to develop this tool. This tool was applied on the study group only. The six-time intervals included the three perioperative stages: the first interval represented the preoperative period, the second interval represented the intraoperative period and the next four intervals represented the postoperative period [over three days after surgery, hospitalization period]. This tool format was prepared in a matrix form that included vertical column representing applicable or not applicable and horizontal row clinical pathway items (as discussed later).

This tool consisted of three phases:

Pre-operative phase; counseling and education of patient for chest physiotherapy, using spirometry, bowel preparation, early mobilization and how to predict common complications with learning to cooperate with nurses. Emphasis on patients to co-operate postoperatively was strongly stressed in spite of the pain and weakness.

Intra-operative phrase: Optimal fluid management, short acting anesthetics, regional analgesia, opioids-sparing anesthesia, small incisions, avoiding drains, maintaining normothermia, venous thrombo-embolism [VTE] prophylaxis and antibiotic prophylaxis were routinely done.

Post-operative phase components: Early oral nutrition, optimal fluid management, multimodal non-opioid analgesia, postoperative nausea and vomiting PONV prophylaxis, stimulation of gut motility, early removal of catheters and drains, early mobilization, chest physiotherapy and using spirometry effectively.

3-Tool three: clinical outcome evaluation: This tool developed by researchers based on reviewing the recent related literature [4]. It was aimed to assess the clinical outcomes for hepatobiliary pancreatic patients three days after surgery and hospitalization period. It was included such as respiratory infection, length of stay in hospital, mortality, fever, admission and readmission to ICU.

ELIGIBILITY:
Inclusion Criteria:

* able to communicate
* Patients without vital failure [renal, hepatic, cardiac].

Exclusion Criteria:

* Past history of other organ cancer
* patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
postoperative pulmonary infection | 6 hours postoperatively, day 1, Day 2, and day 3
  Presence of 3 of the following: tachypnea more than 30/min, expectoration, and hypoxia, respiratory distress

CONTACTS AND LOCATIONS:
Overall Officials: Ayman AM Abouglala, Principal Investigator — Assiut University
Locations (1):
- Faculty of medicine - Assiut university, Asyut, Egypt